CLINICAL TRIAL: NCT03773549
Title: A Virtual Reality Study of Cognitive Biases in Body Dysmorphic Disorder
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, Chief of Psychology, Massachusetts General Hospital
Other Study IDs: 2018P001894
Record Dates: First submitted 2018-12-06; First posted 2018-12-12 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Body Dysmorphic Disorders; Healthy
MeSH Terms: conditions — Body Dysmorphic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Body dysmorphic disorder: Meet DSM-5 criteria for principal body dysmorphic disorder, assessed via the Structured Clinical Interview for the DSM-V Axis I Disorders (SCID)
  Interventions: Other: Virtual reality experience
- Healthy control: Individuals who do not have a current psychiatric diagnosis, assessed via the Mini-International Neuropsychiatric Interview (MINI)
  Interventions: Other: Virtual reality experience

INTERVENTIONS:
Other: Virtual reality experience — Expose all participants (healthy and control) to virtual reality videos while collecting reactivity and self-report outcome measures.

SUMMARY:
Previous research shows that individuals with Body Dysmorphic Disorder (BDD) misinterpret ambiguous social information in a negative and threatening manner. These erroneous threat appraisals are thought to maintain disorder symptomatology and psychosocial impairment by reinforcing individuals' distorted self-image and ideas of social undesirability. Thus, maladaptive interpretation biases represent an important treatment target for this population; however, existing bias assessments and modification protocols are limited by the hypothetical and distal nature of scenarios and do not capture momentary experiential threat processes. The proposed study seeks to test virtual reality (VR) technology as a novel, in vivo means of eliciting, identifying, and measuring threat interpretation biases in a clinical sample to better understand the fear/threat structure activated during social interactions in BDD. Findings have the potential to enhance our understanding of disorder maintenance and identify more nuanced treatment targets. This study represents a critical first step in the long-term goal of harnessing VR gaming technology to supercharge existing treatment approaches for this debilitating illness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+,
* Fluent in English,
* Meet DSM-5 criteria for principal BDD (BDD group) or no other current psychiatric diagnosis (HC group; assessed via clinical interview).

Exclusion Criteria:

* Lifetime psychosis; current bipolar disorder in acute or hypomanic episode; current severe substance use disorder; acute, active suicidal ideation
* Intellectual disability or cognitive impairment that would interfere with participation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with either body dysmorphic disorder or no current psychiatric illness.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Reactivity/arousal of heart rate (HR) during during VR socially ambiguous scenarios | Day 1
  Assessed by using iMotions software to measure heart rate (HR) while watching the virtual reality scenes. We hypothesize that compared to healthy controls, participants with BDD will show greater reactivity/arousal via HR measurements for these socially ambiguous scenarios.
Reactivity/arousal of galvanic skin conductance (GSC) during VR socially ambiguous scenarios | Day 1
  Assessed by using to iMotions software to measure galvanic skin conductance (GSC) while watching the virtual reality scenes. We hypothesize that compared to healthy controls, participants with BDD will show greater reactivity/arousal via GSC measurements for these socially ambiguous scenarios.
Distress ratings | Day 1
  Measured using a brief Likert scale self-report form (author-created distress rating questionnaire) to assess distress, threat, urge to check appearance, and urge to avoid the situation. Ratings will be measured 0-10, with 0 indicating no distress, threat, or urge to check appearance/situation and 10 indicating extreme distress, threat, or urge to check appearance/situation. A maximum score of 40 (a score of 10 on all 4 questions, summed) would indicate extreme distress, while a minimum score of 0 would indicate no distress. Higher scores would indicate greater reactivity.
  We hypothesize that individuals with BDD will score higher on distress ratings than healthy individuals.
Social and appearance-related interpretation biases | Day 1
  We will use the Word-Sentence Association Paradigm (WSAP-BDD) to assess automatic BDD-related threat biases. Participants see ambiguous appearance and/or social sentences paired with a negative/threat and positive/benign interpretation words. Participants rate how related the word and the sentence are; ratings are summed to create "threat" and "benign" subscales. We will also use the Interpretation Questionnaire (IQ) to measure interpretations of everyday situations.
  We hypothesize that compared to healthy controls, BDD participants will show greater endorsement of threat interpretations and lower endorsement of benign interpretations than healthy controls for these interpretation bias measures.
In vivo interpretations | Day 1
  Participants will be presented with two statements for each video exposure; one that articulates a "healthier" benign interpretation and one that articulates a "BDD" interpretation. They will be asked to rate each of the statements for each video.
  We hypothesize that participants with BDD will score higher on BDD interpretations than healthy controls, and that healthy controls will score higher on healthy interpretations than BDD participants.
Correlation of interpretation bias measures | Day 1
  We will look at the correlation between the Word-Sentence Association Paradigm (WSAP-BDD) and the Interpretation Questionnaire (IQ), both established measures of interpretation biases, with our own in vivo bias assessments following the socially ambiguous situations.
  We hypothesize that scores on the previously established WSAP-BDD and IQ will correlate with interpretations on the in vivo bias assessment measures.

SECONDARY OUTCOMES:
Exploratory investigation of acceptability and presence for future treatment using virtual reality methodology | Day 1
  Measured using a brief Likert scale self-report form (author-created measures of acceptability and presence questionnaire) to assess the acceptability of VR technology and presence in VR environment. Ratings will be measured 0-10, with scores of 0 indicating that the participant was not at all engaged with or present in the scenario and that the environment did not at all feel realistic or similar to the real world. Scores of 10 indicate that the participant was completely engaged with or present in the scenario and that the environment felt very realistic or similar to the real world. A maximum score of 50 (a score of 10 on all 5 questions, summed) would indicate complete engagement and high acceptability, while a minimum score of 0 would indicate that the environment was not at all realistic or engaging. Higher scores would show promising future directions for the use of virtual reality technology in this area of research.
Exploratory investigation for future treatment using virtual reality methodology using participant interpretations and feedback on the saliency of the different social contexts. | Day 1
  Measured through a series of open-ended questions regarding particular aspects of the scenes, which were the most/least provocative and realistic, and any alternate interpretations of the ambiguous situations. The open-ended questions are meant to improve future iterations of this work, as the next step will hopefully be a treatment trial.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, Ph.D, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States